CLINICAL TRIAL: NCT02816411
Title: Effects of Protein Supplementation on Skeletal Muscle Regeneration and Healing Process Following Exercise-induced Aseptic Injury
Brief Title: Protein Supplementation and Skeletal Muscle Healing Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PROTEIN-MUSCLEINJURY-2014
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-07

CONDITIONS: Skeletal Muscle Damage; Exercise-induced Aseptic Inflammation; Skeletal Muscle Performance; Intracellular Signaling in Skeletal Muscle; Proteasome Activation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protein (Experimental): Milk protein isolate supplementation: orally, 20g of protein immediately post-exercise and then 20g every 3h on 3 occasions (+3, +6, +9), on the exercise day. The remaining 8 days, 20g daily with breakfast.
  Interventions: Dietary Supplement: Milk protein isolate
- Placebo (Active Comparator): Placebo administration: orally 500 ml, immediately post-exercise as well as at +3, +6 and +9 hours, on the exercise day. The remaining 8 days, 500 ml daily with breakfast.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Milk protein isolate — Milk protein isolate in a powder form consisted of 80% casein and 20% whey protein. 20g were diluted into 500 ml water.
  Placebo consisted of 365 ml water, 125 ml sugar-free cordial and 2g of low-calorie glucose/dextrose powder.
  Arms: Protein
Dietary Supplement: Placebo — 500 mL drink that contained water (375 mL), sugar-free cordial (125 mL) and 2 g of low-calorie glucose/dextrose powder.
  Arms: Placebo

SUMMARY:
In this study the investigators utilized protein supplementation over an 8-day period following eccentric exercise-induced muscle damage in order to test the initial hypotheses : i) protein supplementation after exercise-induced muscle injury affects exercise-induced aseptic inflammation and muscle performance.

DETAILED DESCRIPTION:
The objective was to examine weather protein supplementation is able to affect the inflammatory response as well as recovery of muscle performance following an intense eccentric exercise protocol. In a double-blind, counterbalanced design, 14 men received either Placebo (PLA) or milk protein isolate (PRO) for 8 consecutive days following a single bout of exercise (300 eccentric contractions at 30 deg/sec). In both conditions, performance was assessed at baseline, immediately post-exercise, 2h post-exercise and daily for 8 consecutive days. Blood samples were collected at baseline, 2h post-exercise and daily for the remaining 8 days. Muscle biopsies from vastus lateralis were collected at baseline as well as at day 2 and day 8 of the post-exercise period.

ELIGIBILITY:
Inclusion Criteria:

* a) recreationally trained as indicated by the maximal oxygen consumption levels (VO2max > 45 ml/kg/min), b) engaged in systematic exercise at least three times per week for > 12 months, c) non-smokers, d) abstained from any vigorous physical activity during the study, e) abstained from consumption of caffeine, alcohol, performance-enhancing or antioxidant supplements, and medications during the study.

Exclusion Criteria:

* a) a recent febrile illness, b) history of muscle lesion, c) lower limb trauma

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in reduced glutathione in blood | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
  Concentration of reduced glutathione in red blood cells
Change in protein carbonyls in serum | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
  Concentration of protein carbonyls
Change in protein carbonyls in muscle | 1h before exercise, 2 days post-exercise, 8 days post-exercise
  Protein carbonyl concentration in quadriceps skeletal muscle group
Change in thiobarbituric acid and reactive substances in serum | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
  Thiobarbituric acid reactive substances concentration in serum
Change in oxidized glutathione in blood | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
  Concentration of oxidized glutathione in red blood cells
Change in total antioxidant capacity in serum | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
  Total antioxidant capacity in serum
Change in catalase activity in serum | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
  Catalase activity in serum
Change in creatine kinase activity in plasma | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
Change in C-reactive protein in plasma | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
Change in white blood cell count in blood | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
Changes in volume and morphological complexity of immune cells | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
Change in neutrophil count in blood | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
Change in glucose concentration in blood | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
Change in insulin concentration in blood | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
Change in testosterone concentration in plasma | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
Change in cytokine concentration in plasma | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
  Measurement of IL-1β, IL-4, IL-6, IL-8, IL-10, TNF-α
Change in adhesion molecule concentration in blood | 1h before exercise, 2h post-exercise, daily for 8 days post-exercise
Change in intracellular signalling proteins in muscle | 1h before exercise, 2 days post-exercise, 8 days post-exercise
  Measurement of phosphorylation levels of mammalian target of rapamycin (mTOR), ribosomal protein S6 (rpS6) and nuclear factor kB (NFkB), and protein expression levels of forkhead box protein O1 (FOXO1), HSP70, and parkin.
Change in proteasome activities in muscle | 1h before exercise, 2 days post-exercise, 8 days post-exercise
  Measurement of LLVY, LSTR and LLE
Change in protein expression level of proteasome subunits | 1h before exercise, 2 days post-exercise, 8 days post-exercise
  Measurement of B1i, B2i, B5i, B5, B1, B2 and α7

SECONDARY OUTCOMES:
Change in muscle function of knee extensor and flexor muscle | 1h before exercise, 5 min post-exercise, 2h post-exercise, daily for 8 days post-exercise
  Assessment of muscle peak and mean torque of knee extensors and flexors on an isokinetic dynamometer at 0, 90 and 180 degrees/sec
Body composition | One day before exercise
  Assessment of percent (%) body mass
Maximal aerobic capacity | One day before exercise
  Assessment of maximal oxygen consumption
Change in dietary intake profile | 1h before exercise, daily for 8 days post-exercise
  Assessment of dietary intake with emphasis on protein consumption

CONTACTS AND LOCATIONS:
Overall Officials: IOANNIS G. FATOUROS, Ph.D., Principal Investigator — UNIVERSITY OF THESSALY, SCHOOL OF PHYSICAL EDUCATION & SPORTS SCIENCES
Locations (1):
- Exercise Biochemistry Laboratory, School of Physical Education & Sports Sciences, University of Thessaly, Karies, Trikala, Greece